CLINICAL TRIAL: NCT02439190
Title: A Single Dose Study to Evaluate the Effect of BMS-986120 on Thrombus Formation in an Ex Vivo Thrombosis Chamber Model in Healthy Subjects
Brief Title: CV004-007 Thrombosis Chamber Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CV004-007
Record Dates: First submitted 2015-04-02; First posted 2015-05-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-04

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — BMS-986120; Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A: BMS-986120 (Active Comparator): BMS-986120 on specified days
  Interventions: Drug: BMS-986120
- Treatment B: Aspirin and Clopidogrel (Active Comparator): Aspirin and Clopidogrel on specified days
  Interventions: Drug: Aspirin; Drug: Clopidogrel

INTERVENTIONS:
Drug: BMS-986120
  Arms: Treatment A: BMS-986120
Drug: Aspirin
  Arms: Treatment B: Aspirin and Clopidogrel
Drug: Clopidogrel
  Arms: Treatment B: Aspirin and Clopidogrel

SUMMARY:
The purpose of this study is to determine whether BMS-986120, aspirin, or aspirin and clopidogrel decrease blood clotting.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs and clinical laboratory determinations
* Body Mass Index (BMI) of 18 to 32 kg/m2 inclusive. BMI = weight (kg)/ [height (m)]2
* Females who are not of childbearing potential (i.e., who are post-menopausal or surgically sterile) and men ages 18 to 65, inclusive
* Azoospermic males and women who are not of child-bearing potential (i.e. are postmenopausal or surgically sterile; see section 3.3.3 for the definition of WOCBP) are exempt from contraceptive requirements. However, women must still undergo pregnancy testing as described in this section

Exclusion Criteria:

* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations beyond what is consistent with the target population
* Any condition that could affect drug absorption
* Other protocol-defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in thrombus area (post-treatment with BMS-986120 vs. pre-treatment) | 2 days

SECONDARY OUTCOMES:
Safety and tolerability of BMS 986120 or aspirin administered with and without clopidogrel based on adverse events,clinical laboratory tests, physical examinations and vital signs per the collection schedule | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Derived] Wilson SJ, Ismat FA, Wang Z, Cerra M, Narayan H, Raftis J, Gray TJ, Connell S, Garonzik S, Ma X, Yang J, Newby DE. PAR4 (Protease-Activated Receptor 4) Antagonism With BMS-986120 Inhibits Human Ex Vivo Thrombus Formation. Arterioscler Thromb Vasc Biol. 2018 Feb;38(2):448-456. doi: 10.1161/ATVBAHA.117.310104. Epub 2017 Dec 21. PMID 29269513
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx